CLINICAL TRIAL: NCT05222503
Title: The Impact of Sensor Technology in Individuals With Knee OA
Brief Title: Impact of Sensor Technology in Knee OA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: OPUM Technologies US LTD (Other)
Collaborators: Shirley Ryan AbilityLab (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00214887
Record Dates: First submitted 2022-01-07; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis; knee; orthotics; remote patient monitoring; wearable technology; brace
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control group: Medial off-loader brace and home exercise program (Active Comparator): The subject will receive a traditional medial off-loader brace and a take-home, self-guided exercise program. The subject will be instructed how to wear the brace. The subject will be instructed to incrementally increase wear time of the brace in the first week to get accustomed to the brace to reach a minimum of 6 hours per day after the first week.
  Interventions: Device: Knee Brace
- 2. Intervention group: Medial off-loader brace with OPUM Digital Knee and Remote Patient Monitoring (Experimental): The same off-loader brace as above but with the ODK sensor will be provided. The subject will be instructed how to wear the brace and sensor. The patient will be instructed to incrementally increase wear time in the first week to get accustomed to the brace to reach a minimum of 6 hours per day after the first week. Using the sensor they will be able to keep track of their exercise frequency, range of motion (ROM), and kinematics in the OPUM app on their mobile phone. Education/resources will also be provided to the subjects via modules in the mobile app. The subjects will be instructed how to use the app as well.
  Patients data will be monitored remotely for 20mins per patient per month in the sensor group. Programs will be updated as necessary based on data.
  Interventions: Device: Knee Brace + OPUM Digital Knee

INTERVENTIONS:
Device: Knee Brace + OPUM Digital Knee — Knee Brace + OPUM Digital Knee
  Arms: 2. Intervention group: Medial off-loader brace with OPUM Digital Knee and Remote Patient Monitoring
Device: Knee Brace — Knee Brace without OPUM Digital Knee
  Arms: Control group: Medial off-loader brace and home exercise program

SUMMARY:
OBJECTIVES:

Physical activity has been established as an important component of rehabilitation for knee osteoarthritis (OA), and is often guided by a physical therapist.(1) Physical therapy for knee OA typically involves 1-3 sessions with a licensed physical therapist per week, for up to 12 weeks. These sessions can take a lot of time and effort for subjects, particularly when travel times are considered. Remote patient monitoring is an emerging treatment method which can help to reduce the need for in-person treatment sessions.

Remote patient monitoring has been tested in subjects after a total knee arthroplasty, and initial results show that subjects find the process motivating and engaging.(2) This process has not been tested in individuals with symptomatic knee OA. Prior studies have shown that personalized internet based programs are effective at improving function in individuals with knee OA(3), but the effectiveness of these programs with remote patient monitoring is unknown.

One example of current wearable technology that can be utilized for remote patient monitoring is the Opum (OPUM) Digital Knee® (ODK) modular orthotic. The ODK utilizes a wearable device in a knee brace which relays real time information back to the subject and physical therapist via their mobile phone. The ODK can provide information about sagittal and frontal plane knee kinematics, sagittal plane knee range of motion, time spent performing various daily activities, time spent exercising, overall load on the knee joint, and progress over time in each of these metrics. This device has been previously tested in subjects after an ACL reconstruction, but has yet to be tested in subjects with knee osteoarthritis.

The objective of this study is to assess the effect of the ODK technology in a medial knee unloader brace with remote patient monitoring on pain, function, and quality of life in individuals with knee OA. This study will contain two groups: A control group receiving a medial unloader brace and a personalized home exercise program, and an intervention group which will receive an ODK in a medial off-loader brace, and a home exercise program with remote patient monitoring.

The hypothesis is that subjects who wear the knee brace with the ODK with remote patient monitoring will have a greater reduction in pain and increase in quality of life than those who receive the brace with a home exercise program.

DETAILED DESCRIPTION:
BACKGROUND:

Knee osteoarthritis (OA) is a significant problem in the adult population. With a prevalence of 10-13% in individuals over age 60,(4) knee OA results in a significant reduction in quality of life and increased economic costs to both the individual with knee OA and the medical system as a whole.

Exercise is a key component of management of knee OA, resulting in decreased pain and increased function.(3) Potential barriers to exercise in subjects with knee OA is lack of motivation or professional support.(5) Both of these barriers can be addressed with remote patient monitoring. Remote patient monitoring will allow a physical therapist to monitor the activity levels and progress of each subject, and make adjustments throughout the duration the rehab program.

Wearable technology has begun to disrupt conventional methods of healthcare delivery. Wearable technology can allow for remote patient monitoring and self monitoring for subjects with OA. The ODK is a novel wearable device which has previously been tested in subjects with anterior cruciate ligament (ACL) reconstructions, but has not yet been tested in individuals with knee OA. The ODK allows for tracking of knee range of motion, frontal plane kinematics, sagittal plane kinematics, exercise progress, time spent walking/standing/sitting/kneeling, and time spent sedentary. These measures can help to provide useful information to the patient on potential mitigating factors in their knee OA and provide real time feedback about joint kinematics.

This study will investigate the effects of the ODK used in a medial off-loader brace with remote patient monitoring. This randomized control trial will have 2 groups: A control group receiving a medial unloader brace and a personalized home exercise program, and an intervention group which will receive an ODK in a medial off-loader brace, and a home exercise program with remote patient monitoring. These subjects will be followed for 12 weeks and assessed for changes in pain, function, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Pain score > 12.5 KOOS
* BMI < 35
* Own a compatible mobile phone?
* Able to operate Bluetooth technology?
* Diagnosis of unilateral femoro-tibial knee OA

Exclusion Criteria:

* History of lower extremity total joint arthroplasty? (in affected knee)
* Current uncontrolled cardiovascular disease?
* Other pathology? Ex: Parkinson's, stroke, multiple sclerosis (MS), amyotrophic lateral sclerosis (ALS), or other knee diseases (Paget, osteonecrosis, etc.)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-07-14 (Estimated)

PRIMARY OUTCOMES:
Pain subscore on the Knee injury and Osteoarthritis Score (KOOS Survey) | 12 weeks from onset of brace wearing
  Measured by the Knee injury and osteoarthritis score subscale (KOOS subscales) as a comparison between both groups of the evolution of pain between Day 0 and Week 12.

SECONDARY OUTCOMES:
Symptoms | 12 weeks from onset of brace wearing
  Measured by the Symptoms Knee injury and osteoarthritis score subscales (KOOS subscales) as a comparison between day 0 and week 12.
Function | 12 weeks from onset of brace wearing
  Measured by the Function Knee injury and osteoarthritis score subscales (KOOS subscales) as a comparison between day 0 and week 12.
Impact of Osteoarthritis on Quality of Life | 12 weeks from onset of brace wearing
  Measured by the Quality of life Knee injury and osteoarthritis score subscales (KOOS subscales) as a comparison between day 0 and week 12.
Quality of life measured using the EQ5D survey | 12 weeks from onset of brace wearing
  Measured via the EQ5D survey as a comparison from day 0 and week 12.
Walking speed | 12 weeks from onset of brace wearing
  Measured using the 10 m walk test: participants are timed as they walk 10m and this walking speed is calculated using (speed = distance/time) in m/s. Done on day 0 and compared to week 12
Walking endurance | 12 weeks from onset of brace wearing
  Measured using 6min walk test: participant walks for 6 minutes and the distance (m) walked is measured. If needed, the number of breaks taken is noted. Test done on day 0 and compared to week 12
Stair negotiation | 12 weeks from onset of brace wearing
  Participants are timed (seconds) as they ascend and descend a flight of stairs. Done on day 0 and after 12 weeks of brace wearing; times are compared.
5 times sit-to-stand | 12 weeks from onset of brace wearing
  Participants are timed (seconds) as they stand from a seated position in a chair and sit back down 5 times. This exercise is timed on day 0 and after 12 weeks of brace wearing; times are compared.
Patient diary | 12 weeks
  Self-reported compliance with brace wearing and exercise program
Digital Knee Data (for intervention group) | 12 weeks
  Activity recorded by the ODK module for the intervention group during the 12 week intervention
Patient satisfaction | At 12-week follow-up visit
  Survey administered after the 12 week intervention that assessed patient satisfaction using questions about likelihood of having surgical treatment in the 12 months that followed the study.
  One question asked if patients were A. More Likely, B. Less Likely, C. Unchanged Another question asked patients to indicate on a scale of 0-100, how likely they were to get surgery where 0=unlikely and 100=very likely.
  Another question that asked whether or not patients would continue to use the program after completion of the study time period.
System Usability Scale (for intervention group) | At 12-week follow-up visit
  A survey administered to get feedback on the user-friendliness of the device and application. With an optional space for additional feedback. Participants' impression of the program are assessed by presenting multiple sentences such as "I found this device easy to use" and asking the participant to rank the statement on a scale of 1 to 5, where 1 = strongly disagree and 5 = strongly agree.
Condition Improvement | At 12-week follow-up visit
  Survey questions addressing perceived change in condition by asking patients to (one question): describe the change in ACTIVITY, LIMITATIONS, SYMPTOMS, EMOTIONS, and OVERALL QUALITY OF LIFE associated with your osteoarthritis condition.
  The answer choices were:
  A. No change (Or condition has gotten worse) B. Almost the same, hardly any change at all C. A little better, but no noticeable change D. Somewhat better, but the change has not made any real difference E. Moderately better, and a slight but noticeable change F. Better and a definite improvement that has made a real and worthwhile difference G. A great deal better and a considerable improvement that has made all the difference
  Another survey question addressing perceived change in condition by indicating their improvement on a scale of 0-100 where 0 = very much worse, 50 = unchanged, and 100 = very much better.
Need for medication to treat osteoarthritis symptoms | At 12-week follow-up visit
  Assessed in the form of a survey question that asked participants to describe the amount of medication they take for their osteoarthritis since the onset of the study.
  The answer choices were: UNCHANGED, STOPPED, DECREASED, INCREASED, N/A

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Jayabalan, MD, PhD, Principal Investigator — Shirley Ryan AbilityLab; Northwestern University Feinberg School of Medicine
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Clin Geriatr Med. 2010 Aug;26(3):355-69. doi: 10.1016/j.cger.2010.03.001. PMID 20699159
- [Result] Bhatia D, Bejarano T, Novo M. Current interventions in the management of knee osteoarthritis. J Pharm Bioallied Sci. 2013 Jan;5(1):30-8. doi: 10.4103/0975-7406.106561. PMID 23559821
- [Result] Ramkumar PN, Haeberle HS, Ramanathan D, Cantrell WA, Navarro SM, Mont MA, Bloomfield M, Patterson BM. Remote Patient Monitoring Using Mobile Health for Total Knee Arthroplasty: Validation of a Wearable and Machine Learning-Based Surveillance Platform. J Arthroplasty. 2019 Oct;34(10):2253-2259. doi: 10.1016/j.arth.2019.05.021. Epub 2019 May 16. PMID 31128890
- [Result] Bosomworth NJ. Exercise and knee osteoarthritis: benefit or hazard? Can Fam Physician. 2009 Sep;55(9):871-8. PMID 19752252
- [Result] Kanavaki AM, Rushton A, Efstathiou N, Alrushud A, Klocke R, Abhishek A, Duda JL. Barriers and facilitators of physical activity in knee and hip osteoarthritis: a systematic review of qualitative evidence. BMJ Open. 2017 Dec 26;7(12):e017042. doi: 10.1136/bmjopen-2017-017042. PMID 29282257